CLINICAL TRIAL: NCT01388361
Title: A Trial Comparing the Efficacy and Safety of Adding Liraglutide Versus Addition of Insulin Aspart With the Largest Meal to Insulin Degludec, Both in Combination With Metformin, in Subjects With Type 2 Diabetes Qualifying for Treatment Intensification (BEGIN™: VICTOZA® ADD-ON)
Brief Title: Comparison of the Efficacy and Safety of Two Intensification Strategies in Subjects With Type 2 Diabetes Inadequately Controlled on Basal Insulin and Metformin
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3948; 2011-001493-25 (EudraCT Number); U1111-1120-2782 (Other: WHO)
Record Dates: First submitted 2011-07-04; First posted 2011-07-06 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Aspart; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IDeg (non-randomised) (Experimental)
  Interventions: Drug: insulin degludec
- IDeg + IAsp (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- IDeg + liraglutide (Experimental)
  Interventions: Drug: insulin degludec; Drug: liraglutide

INTERVENTIONS:
Drug: insulin degludec — Injected s.c. (under the skin) once daily. The doses will be individually adjusted
Drug: insulin aspart — Injected s.c. (under the skin) once daily. The doses will be individually adjusted.
  Arms: IDeg + IAsp
Drug: liraglutide — Injected s.c. (under the skin) once daily. The doses will be individually adjusted.
  Arms: IDeg + liraglutide

SUMMARY:
This trial is conducted in Europe and North America. The aim of this trial is to compare the efficacy and safety of adding liraglutide versus addition of insulin aspart with the largest meal to insulin degludec in subjects with type 2 diabetes.

Eligible subjects with an HbA1c equal to or above 7% at end of treatment in NN1250-3643 (NCT01193309) trial will be randomised to receive treatment intensification while subjects with an HbA1c below 7% at end of treatment in NN1250-3643 (NCT01193309) may continue to receive insulin degludec treatment. Subjects are to continue their pre-trial metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject).
* The subject must have completed the end of treatment visit of NN1250-3643 with Insulin degludec once daily + metformin.
* Ability and willingness to adhere to the protocol including self measurement of plasma glucose according to the protocol

Exclusion Criteria:

* Participated in NN1250-3643 and treated with insulin glargine
* Previous treatment with glucacon like peptide (GLP-1) receptor agonists (e.g. exenatide, liraglutide)
* Impaired liver function, defined as alanine aminotransferase (ALAT) 2.5 times the upper limit of normal at end of treatment in NN1250-3643
* Impaired renal function defined as serum-creatinine = 125 µmol/l (= 1.4 mg/dl) for males and = 110 µmol/L (= 1.3 mg/dl) for females or according to local label for metformin [For France: glomerular filtration rate below 60 ml/min, calculated by the Cockroft & Gault formula] at end of treatment in NN1250-3643.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (118):
- United States (47):
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, National City, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Tarzana, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, North East, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Melrose Park, Pennsylvania
  - Novo Nordisk Investigational Site, Upper Saint Clair, Pennsylvania
  - Novo Nordisk Investigational Site, East Providence, Rhode Island
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Austria (3):
  - Novo Nordisk Investigational Site, Feldkirch
  - Novo Nordisk Investigational Site, Vienna
  - Novo Nordisk Investigational Site, Wolfsberg
- Belgium (4):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Liège
- Canada (14):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Coquitlam, British Columbia
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Scarborough Village, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Québec, Quebec
  - Novo Nordisk Investigational Site, Saint Romuald, Quebec
  - Novo Nordisk Investigational Site, Saint-Marc-des-Carrieres, Quebec
- Czechia (4):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prague
- Denmark (6):
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Hillerød
  - Novo Nordisk Investigational Site, Holbæk
  - Novo Nordisk Investigational Site, København S
  - Novo Nordisk Investigational Site, Odense
  - Novo Nordisk Investigational Site, Silkeborg
- Finland (6):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Joensuu
  - Novo Nordisk Investigational Site, Kerava
  - Novo Nordisk Investigational Site, Lohja
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Tampere
- France (4):
  - Novo Nordisk Investigational Site, Montigny-lès-Metz
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (12):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Rehburg-Loccum
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Speyer
- Norway (8):
  - Novo Nordisk Investigational Site, Ålesund
  - Novo Nordisk Investigational Site, Bekkestua
  - Novo Nordisk Investigational Site, Elverum
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- Serbia (4):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Spain (6):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Antequera
  - Novo Nordisk Investigational Site, Ferrol
  - Novo Nordisk Investigational Site, Inca
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Seville

REFERENCES:
- [Result] Mathieu C, Rodbard HW, Cariou B, Handelsman Y, Philis-Tsimikas A, Ocampo Francisco AM, Rana A, Zinman B; BEGIN: VICTOZA ADD-ON (NN1250-3948) study group. A comparison of adding liraglutide versus a single daily dose of insulin aspart to insulin degludec in subjects with type 2 diabetes (BEGIN: VICTOZA ADD-ON). Diabetes Obes Metab. 2014 Jul;16(7):636-44. doi: 10.1111/dom.12262. Epub 2014 Feb 11. PMID 24443830
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 119 sites in 12 countries: Austria (4), Belgium (4), Canada (15), Czech Republic (4), Denmark (6), Finland (6), France (4), Germany (12), Norway (6), Serbia (5), Spain (7) and United States (46). These sites enrolled subjects in the randomised or non-randomised arms of the trial.
Pre-assignment Details: Subjects treated with Insulin degludec (IDeg) once daily (OD) + metformin in trial NN1250-3643 (NCT01193309) were eligible for this trial. Eligible subjects with an HbA1c >/=7.0% at the end of 3643 trial were qualified to enter the extension trial 3948 and be randomised to add either liraglutide/insulin aspart to their prior IDeg + Met treatment.
Groups:
- IDeg: This non-randomised arm consisted of subjects treated with IDeg + metformin who achieved the target glycosylated haemoglobin (HbA1c) < 7.0 % at the end of treatment in NN1250-3643. Subjects were treated with once-daily subcutaneous administration of IDeg 100 U/mL prefilled pen along with stable and pre-trial dose of oral antidiabetic drug metformin for 26-weeks. These subjects continued on IDeg + metformin to assess the treatment regimen's ability to sustain long term glycaemic control. No comparisons of endpoints were made between the non-randomised and randomised treatment arms.
- IDeg + Liraglutide: All subjects in this arm were randomised to once-daily subcutaneous administration of IDeg 100 U/mL in a prefilled pen along with once-daily subcutaneous administration of liraglutide (6 mg/mL) in a prefilled pen for 26 weeks of treatment. Subjects continued their oral antidiabetic drug metformin at a stable, pre-trial dose throughout the trial period.
- IDeg + IAsp OD: Subjects in this arm were randomised to once-daily subcutaneous administration of IDeg 100 U/mL in prefilled pen along with once-daily subcutaneous administration of insulin aspart (IAsp)100 U/mL in a FlexPen® administered just before the largest meal for 26 weeks of treatment. Subjects continued their oral antidiabetic drug metformin at a stable, pre-trial dose throughout the trial period.
Period: Overall Study
Arm/Group | IDeg | IDeg + Liraglutide | IDeg + IAsp OD
Started | 236 | 88 | 89
Exposed | 234 (Two subjects withdrew prior to exposure to IDeg during NN1250-3948) | 87 (One subject withdrew prior to exposure to trial drug.) | 86 (Three subjects withdrew prior to exposure to trial drug.)
Completed | 224 | 76 | 75
Not Completed | 12 | 12 | 14
Not completed — Adverse Event | 0 | 5 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal criteria | 12 | 7 | 10
Not completed — Unclassified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised patients except for 7 subjects (2 subjects with IDeg+ liraglutide; 5 subjects with IDeg+IAsp arm) fasting plasma glucose (FPG) values were missing at baseline. Non-randomised set (NAS) included all non-randomised subjects, the FPG values were missing for 10 subjects at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg | IDeg + Liraglutide | IDeg + IAsp OD | Total
Number analyzed (Participants) | 236 | 88 | 89 | 413
Age, Continuous [Mean (Standard Deviation); unit: years] — Non-randomised population.
  years | 61.9 (9.3) | NA (NA) — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | NA (NA) — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | 61.9 (9.3)
Age, Continuous [Mean (Standard Deviation); unit: years] — Randomised population.
  years | NA (NA) — Values available in the previous row, baseline values for non-randomised arm IDeg. | 61.1 (9.5) | 60.9 (8.8) | 61.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Non-randomised population.
  Participants
    Female | 90 | NA — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | NA — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | 146 | NA — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | NA — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants] — Randomised population.
  Participants
    Female | NA — Values available in the previous row, baseline values for non-randomised arm IDeg. | 25 | 36 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — Values available in the previous row, baseline values for non-randomised arm IDeg. | 63 | 53 | NA — Total not calculated because data are not available (NA) in one or more arms.
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] — Non-randomised population.
  percentage of glycosylated haemoglobin | 6.4 (0.4) | NA (NA) — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | NA (NA) — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | 6.4 (0.4)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] — Randomised population.
  percentage of glycosylated haemoglobin | NA (NA) — Values available in the previous row, baseline values for non-randomised arm IDeg. | 7.7 (0.6) | 7.7 (0.8) | 7.7 (0.7)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — Non-randomised population.
  mmol/L | 6.7 (1.8) | NA (NA) — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | NA (NA) — Values available in the next row, baseline values for IDeg + Liraglutide vs. IDeg + IAsp OD. | 6.7 (1.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — Randomised population.
  mmol/L | NA (NA) — Values available in the previous row, baseline values for non-randomised arm IDeg. | 6.4 (2.4) | 6.1 (1.7) | 6.3 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (%) (Glycosylated Haemoglobin)
Description: Values for change in HbA1c from baseline to 26 weeks of treatment period.
Time Frame: week 0, week 26
Population: The FAS and NAS included all randomised and non-randomised subjects respectively, and missing data was imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg | IDeg + Liraglutide | IDeg + IAsp OD
Number analyzed (Participants) | 236 | 88 | 89
percentage of glycosylated haemoglobin | 0.10 (0.40) | -0.74 (0.73) | -0.39 (0.72)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Values for change in FPG in mmol/L from baseline to week 26 of randomised period.
Time Frame: week 0, week 26
Population: Both sets of FAS and NAS included all randomised and non-randomised subjects in the treatment period. The FPG values were missing for 7 subjects in FAS (2 subjects with IDeg+ liraglutide; 5 subjects with IDeg+IAsp arm) and 10 subjects in NAS for IDeg arm at baseline. The missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg | IDeg + Liraglutide | IDeg + IAsp OD
Number analyzed (Participants) | 226 | 86 | 84
mmol/L | -1.23 (2.03) | -0.14 (2.52) | -0.04 (2.84)

3. Secondary Outcome: Change From Baseline in Body Weight
Description: Corresponds to the values of change in body weight in kilograms from baseline to week 26.
Time Frame: week 0, week 26
Population: Both sets of FAS and NAS included all randomised and non-randomised subjects in the treatment period and missing data was imputed using LOCF. At baseline, the body weight values were missing for 1 subject in IDeg + Liraglutide arm from FAS and 3 subjects in NAS for IDeg arm.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDeg | IDeg + Liraglutide | IDeg + IAsp OD
Number analyzed (Participants) | 233 | 87 | 89
kg | 0.1 (2.7) | -1.0 (1.3) | 0.3 (0.9)

4. Secondary Outcome: Number of Severe and Minor Treatment Emergent Hypoglycaemic Episodes
Description: Corresponds to number of treatment emergent hypoglycaemic events from onset on or after the first day of exposure to investigational product and no later than 7 days after last exposure to investigational product. Confirmed hypoglycaemia was defined as the pool of severe hypoglycaemic episodes and minor episodes with a plasma glucose (PG) value < 3.1 mmol/L (56 mg/dL).
Time Frame: Onset on or after the first day of exposure to investigational product for 26 weeks of treatment period and no later than 7 days after last exposure to investigational product.
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator
Measure: Number; unit: events
Arm/Group | IDeg | IDeg + Liraglutide | IDeg + IAsp OD
Number analyzed (Participants) | 236 | 87 | 86
events
  Confirmed(severe+minor) | 313 | 40 | 330
  Severe | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected during 26 week treatment period + 7 days follow up.
Description: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg | IDeg + Liraglutide | IDeg + IAsp OD
Serious Adverse Events (participants affected / at risk) | 11/236 | 4/87 | 5/86
Other Adverse Events (participants affected / at risk) | 64/236 | 40/87 | 18/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=236) | IDeg + Liraglutide (N=87) | IDeg + IAsp OD (N=86)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=236) | IDeg + Liraglutide (N=87) | IDeg + IAsp OD (N=86)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 9 (12) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 18 (25) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (5) | 0 (0)
Bronchitis (Infections and infestations) | 13 (14) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 43 (54) | 9 (11) | 11 (12)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 4 (5) | 3 (3)
Lipase increased (Investigations) | 0 (0) | 6 (7) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.